CLINICAL TRIAL: NCT04458831
Title: A Prospective, Non-interventional, Multinational, Observational Study With Isatuximab in Patients With Relapsed and/or Refractory Multiple Myeloma (RRMM)
Acronym: IONA-MM
Status: Active, not recruiting | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS16577
Record Dates: First submitted 2020-06-25; First posted 2020-07-07 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — isatuximab; pomalidomide; Dexamethasone; carfilzomib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Patients with multiple myeloma (MM) and are considered as RRMM according to the International Myeloma Working Group (IMWG) criteria
  Interventions: Drug: isatuximab SAR650984; Drug: Pomalidomide; Drug: Dexamethasone; Drug: Carfilzomib

INTERVENTIONS:
Drug: isatuximab SAR650984 — Pharmaceutical form: solution for infusion
  Route of administration: intravenous
  Other Names: Sarclisa
Drug: Pomalidomide — Pharmaceutical form: oral
  Other Names: Pomalyst
Drug: Dexamethasone — Pharmaceutical form: oral
Drug: Carfilzomib — Pharmaceutical form: solution for infusion

SUMMARY:
Primary Objective:

To assess the effectiveness, in terms of overall response rate (ORR) of isatuximab patients with RRMM in routine clinical practice, within 12 months

To assess other effectiveness parameters such as progression free survival (PFS), PFS rate (PFSR), duration of response (DoR), time to response, time and intent to first subsequent therapy, rate of very good partial response or better, rate of complete response (CR) or better of isatuximab patients with RRMM in routine clinical practice

To assess the profile of patients (demographic, disease characteristics, comorbidities and prior MM treatment history) who are treated with isatuximab in routine clinical practice

To describe safety of isatuximab in routine clinical practice (based on adverse event [AE] reporting)

To assess quality of life (QoL) using the European Organization for Research and Treatment of Cancer (EORTC) 30 item core questionnaire (QLQ C30) and the accompanying 20 item myeloma questionnaire module (QLQ MY20)

Secondary Objective:

Not applicable

DETAILED DESCRIPTION:
Duration per participant is 2.5 years

ELIGIBILITY:
* Age ≥18 years or country's legal age of majority if the legal age is >18 years old at the time of enrollment
* Patients with RRMM who have at least one prior line of therapy
* Patients for whom the treating physician has made the decision to initiate isatuximab per routine practice and independently of the purpose of the study; for retrospectively enrolled patients, exposure to isatuximab treatment for a maximum of three months prior to study enrollment
* Able to understand and complete the study-related questionnaires
* Patient must have given signed informed consent prior to study start. For retrospectively enrolled patients who are deceased at the date of enrollment into the study, a waiver of consent will be required; patients who have started and stopped treatment or whose treatment is still ongoing at ICF are eligible

Most important exclusion criteria for potential participants:

* Patients who are receiving isatuximab for an indication other than RRMM
* Patients who have received any other investigational drug or prohibited therapy for this study within 28 days or five half-lives from randomization, whichever is longer
* Patients having contraindication to the isatuximab summary of product characteristics (SMPC) or package insert (PI)
* Patients having contraindications as noted in the drug-specific local isatuximab SMPC/PI of combination drugs
* Any country-related specific regulation that would prevent the patient from entering the study

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial. Further eligibility criteria might apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The source population for this study will be patients with a diagnosis of RRMM recruited from participating sites in Asia, Europe, Latin America, and North America. The study will aim to enroll up to approximately 640 adult patients with a recorded diagnosis of RRMM from up to 150 sites. A subset of patients from sites, limited to the US and UK only, will be recruited (up to 100 patients out of 640), for enrichment by leveraging existing electronic medical record (EMR) technologies coupled with the electronic case report forms (eCRFs).
Sampling Method: Probability Sample
Enrollment: 583 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2026-02-23 (Estimated); Study Completion 2026-02-23 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 12 months
  The proportion of patients with stringent complete response (sCR), complete response (CR), very good partial response (VGPR), and partial response (PR) as best overall response assessed by investigator using the IMWG response criteria
Progression free survival (PFS) | Up to 30 months
  Time from isatuximab start date to the date of first documentation of progressive disease (PD) (as determined by the investigator) or the date of death from any cause, whichever comes first.
Progression free survival rate (PFSR) | up to 18 months
  The proportion of patients who do not progress and are alive at a specific time intervals
Duration of response (DoR) | Up to 30 months
  Time from the date of the first response for patients achieving partial response (PR) 4 or better (PR, VGPR, CR, or sCR) to the date of first documented PD (as determined by Investigator using the IMWG response criteria) or death, whichever happens first.
Time to response (TTR) | Up to 30 months
  Defined as the time between isatuximab start date and the onset of first response for patients achieving PR or better (sCR, CR, VGPR, or PR) assessed by investigator using the IMWG response criteria
Time to first subsequent anti-myeloma therapy | Up to 30 months
  Time from the initiation of isatuximab until the start of subsequent therapy or death.
Rate of very good partial response or better | 12 months
  Comprising VGPR, CR, and sCR within 12 months
Rate of complete response (CR) or better | 12 months
  Comprising CR and sCR responses within 12 months
Number of Participants with Adverse events | Up to 1 month after the end of treatment
  Adverse events (AE) including treatment emergent adverse events (TEAE), serious adverse events (SAE) and adverse events of special interest (AESIs) according to the following parameters: infusion associated reactions (IARs), pregnancy in a patient (or partner of a patient), symptomatic overdose, occurrence of a second primary malignancy, and/or neutropenia. TEAEs are defined as AEs that develop, worsen (according to the Investigator opinion), or become serious during the TEAE period infusion
Change from Baseline in the European Organization for Research and Treatment of Cancer (EORTC) Disease-Related Symptom Scales of the Quality of Life 30 item core questionnaire (QLQ-C30) | through end of treatment (up to approximately 2 years)
  EORTC QLQ-MY20 standardized scores: The EORTC QLQ-C30 is a brief self- or interviewer-administered patient-reported survey. This 30-item questionnaire measures the following domains: 1) global health status/QoL; 2) functional scales including physical, role, emotional, cognitive, and social functioning; and 3) symptom scales/items related to fatigue, nausea and vomiting, pain, dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial impact.
Change from Baseline in the EORTC Multiple Myeloma Specific Quality of Life 20 item questionnaire (QLQ MY20) | through end of treatment (up to approximately 2 years)
  EORTC QLQ-C30 standardized scores: The EORTC QLQ-MY20 is a validated, self -administered instrument to assess QoL in persons with MM. This 20-item questionnaire measures the following domains: symptom scales, including disease symptoms (6 items) and symptoms related to side effects of treatment (10 items); function scale and future perspective (3 items); and body image (1 item).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (129):
- United States (24):
  - University of Arkansas Medical Sciences Site Number : 8400021, Little Rock, Arkansas
  - St. Joseph Heritage Healthcare Site Number : 8400008, Fullerton, California
  - University of California San Francisco (PARENT) Site Number : 8400009, San Francisco, California
  - Holy Cross Hospital Site Number : 8400030, Fort Lauderdale, Florida
  - GenesisCare Site Number : 8400007, Jacksonville, Florida
  - Watson Clinic Cancer and Research Center Site Number : 8400023, Lakeland, Florida
  - Millennium Oncology Site Number : 8400025, Pembroke Pines, Florida
  - Comprehensive Hematology Oncology Site Number : 8400026, St. Petersburg, Florida
  - Central Care Cancer Center Site Number : 8400019, Garden City, Kansas
  - Central Maine Medical Center Site Number : 8400031, Lewiston, Maine
  - Michigan Center of Medical Research Site Number : 8400010, Farmington Hills, Michigan
  - Central Care Cancer Center Site Number : 8400006, Garden City, Missouri
  - AMR Kansas City Site Number : 8400016, Kansas City, Missouri
  - Regional Cancer Care Associates, LLC - Freehold Division Site Number : 8400017, Freehold, New Jersey
  - Regional Cancer Care Associates Site Number : 8400024, Howell Township, New Jersey
  - Regional Cancer Care Associates - Little Silver Division Site Number : 8400018, Little Silver, New Jersey
  - Novant Health Forsyth Medical Center Site Number : 8400028, Winston-Salem, North Carolina
  - Hematology & Oncology Associates Site Number : 8400015, Canton, Ohio
  - Tri County Hematology & Oncology Associates, Inc Site Number : 8400012, Massillon, Ohio
  - Charleston Hematology Oncology Associates, PA Site Number : 8400020, Charleston, South Carolina
  - Prisma Health - Eastside Office Site Number : 8400011, Greenville, South Carolina
  - Prairie Lakes Health Care System, Inc Site Number : 8400002, Watertown, South Dakota
  - MD Anderson Cancer Center Site Number : 8400013, Houston, Texas
  - Renovatio Clinical Site Number : 8400004, The Woodlands, Texas
- Argentina (5):
  - Investigational Site Number : 0320001, Ciudad Autonoma Buenos Aires, Buenos Aires
  - Investigational Site Number : 0320006, Pilar, Buenos Aires
  - Investigational Site Number : 0320004, Buenos Aires
  - Investigational Site Number : 0320005, Córdoba
  - Investigational Site Number : 0320002, Córdoba
- LKH Steyr - Investigational Site Number : 0400002, Steyr, Austria
- Belgium (2):
  - Institut Jules Bordet - Investigational Site Number : 0560001, Anderlecht
  - AZ Nikolaas - Investigational Site Number : 0560002, Sint-Niklaas
- China (2):
  - Investigational Site Number : 1560002, Guangzhou
  - Investigational Site Number : 1560001, Shenzhen
- France (15):
  - Centre Hospitalier Victor Dupouy - Investigational Site Number : 2500007, Argenteuil
  - Investigational Site Number : 2500017, Cahors
  - Centre Hospitalier Metropole Savoie - Investigational Site Number : 2500006, Chambéry
  - Clinique Louis Pasteur, Maison Médicale - Investigational Site Number : 2500012, Essey-lès-Nancy
  - Centre Hospitalier Le Mans - Investigational Site Number : 2500015, Le Mans
  - Investigational Site Number : 2500013, Lille
  - Investigational Site Number : 2500004, Montpellier
  - Investigational Site Number : 2500009, Pessac
  - CHU Poitiers - Hôpital la Milétrie - Investigational Site Number : 2500008, Poitiers
  - CHU Reims - Hôpital Robert Debré - Investigational Site Number : 2500010, Reims
  - Investigational Site Number : 2500001, Rouen
  - Investigational Site Number : 2500005, Saint-Priest-en-Jarez
  - Investigational Site Number : 2500014, Saint-Quentin
  - Investigational Site Number : 2500016, Tarbes
  - Investigational Site Number : 2500011, Vannes
- Germany (28):
  - Investigational Site Number : 2760016, Aschaffenburg
  - Investigational Site Number : 2760020, Bamberg
  - Investigational Site Number : 2760018, Bayreuth
  - Investigational Site Number : 2760003, Berlin
  - Investigational Site Number : 2760041, Berlin
  - Praxis am Volkspark - Investigational Site Number : 2760009, Berlin
  - Investigational Site Number : 2760022, Berlin
  - MV Zentrum für Onkologie und Hämatologie - Investigational Site Number : 2760034, Cologne
  - Investigational Site Number : 2760007, Donauwörth
  - GEFOS Gesellschaft f. onkologische Studien -Investigational Site Number : 2760001, Dortmund
  - Investigational Site Number : 2760002, Dresden
  - Investigational Site Number : 2760035, Dresden
  - Investigational Site Number : 2760037, Frankfurt
  - Onkologische Gemeinschaftspraxis am Bethanien-Krankenhaus - Investigational Site Number : 2760010, Frankfurt am Main
  - Investigational Site Number : 2760012, Hanover
  - Investigational Site Number : 2760013, Herrsching am Ammersee
  - Klinikum Kulmbach mit Fachklinik Stadtsteinach - Investigational Site Number : 2760026, Kulmbach
  - Investigational Site Number : 2760008, Leipzig
  - Philipps-Universitat Marburg, Klinic fur Innere Medizin -Investigational Site Number : 2760038, Marburg
  - Klinikum Schwaebisch Gmuend - Investigational Site Number : 2760042, Mutlangen
  - Investigational Site Number : 2760006, München
  - Dietrich-Bonhoeffer-Klinikum - Investigational Site Number : 2760044, Neubrandenburg
  - Investigational Site Number : 2760021, Oldenburg
  - Investigational Site Number : 2760036, Oldenburg
  - Klinikum Ernst von Bergmann gGmbH -Investigational Site Number : 2760039, Potsdam
  - Investigational Site Number : 2760040, Stolberg
  - Investigational Site Number : 2760031, Weilheim
  - Investigational Site Number : 2760019, Würzburg
- Investigational Site Number : 3000005, Piraeus, Greece
- Investigational Site Number : 3440001, Hong Kong, Hong Kong
- Italy (11):
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia - Investigational Site Number : 3800009, Rome, Roma
  - Azienda Ospedaliera Universitaria Policlinico Umberto I - Investigational Site Number : 3800002, Rome, Roma
  - Investigational Site Number : 3800006, Bari
  - Istituto di Ematologia e Oncologia Medica - Investigational Site Number : 3800005, Bologna
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia - Investigational Site Number : 3800007, Brescia
  - Investigational Site Number : 3800003, Milan
  - Azienda Ospedaliera Universitaria "Federico II"-Investigational Site Number : 3800001, Napoli
  - Investigational Site Number : 3800008, Novara
  - Investigational Site Number : 3800013, Pavia
  - Investigational Site Number : 3800004, Trento
  - Investigational Site Number : 3800010, Treviso
- Japan (11):
  - Investigational Site Number : 3920012, Sapporo, Hokkaido
  - Investigational Site Number : 3920009, Osaka, Osaka
  - Investigational Site Number : 3920003, Sunto-gun, Shizuoka
  - Investigational Site Number : 3920004, Minato-ku, Tokyo
  - Investigational Site Number : 3920010, Fukuoka
  - Investigational Site Number : 3920013, Minatoku
  - Investigational Site Number : 3920005, Okayama
  - Investigational Site Number : 3920014, Osakasayama-shi
  - Investigational Site Number : 3920008, Shibukawa-shi
  - Investigational Site Number : 3920011, Suwa-shi
  - Investigational Site Number : 3920001, Yamagata
- Investigational Site Number : 4140001, Kuwait City, Kuwait
- Albert Schweitzer Ziekenhuis - Investigational Site Number : 5820001, Dordrecht, Netherlands
- Puerto Rico (2):
  - Puerto Rico Medical Research Center, LLC Site Number : 8400001, Hato Rey
  - Auxilio Mutuo Cancer Center Site Number : 8400029, San Juan
- Investigational Site Number : 6430006, Volgograd, Russia
- Saudi Arabia (4):
  - Investigational Site Number : 6820005, Jeddah
  - Investigational Site Number : 6820004, Jeddah
  - Investigational Site Number : 6820001, Khobar
  - Investigational Site Number : 6820002, Riyadh
- Spain (8):
  - Hospital Universitari Son Espases - Investigational Site Number : 7240003, Palma de Mallorca, Balearic Islands
  - Complejo Asistencial Universitario de Leon Altos de Nava s/n. -Investigational Site Number : 7240005, León, León
  - Hospital Regional Universitario de Malaga Hospital Regional Universitario de Malaga - Investigational Site Number : 7240006, Málaga, Málaga
  - Hospital Universitario de Navarra - Investigational Site Number : 7240009, Pamplona, Navarre
  - Hospital Universitario Virgen de la Nieves - Investigational Site Number : 7240010, Granada
  - Complejo Hospitalario Universitario de Pontevedra - Investigational Site Number : 7240011, Pontevedra
  - omplejo Hospitalario Universitario de Canarias - Investigational Site Number : 7240007, San Cristóbal de La Laguna
  - Investigational Site Number : 7240004, Toledo
- Switzerland (3):
  - Kantonsspital Baden AG - Investigational Site Number : 5760003, Baden
  - Investigational Site Number : 5760001, Bern
  - Stadtspital Triemli - Investigational Site Number : 5760002, Zurich
- Taiwan (2):
  - Investigational Site Number : 1580002, Kaohsiung City
  - Investigational Site Number : 1580001, Taipei
- United Arab Emirates (2):
  - Investigational Site Number : 7840002, Abu Dhabi
  - Investigational Site Number : 7840001, Abu Dhabi
- United Kingdom (4):
  - Investigational Site Number : 8260002, Nottingham, Nottinghamshire
  - Investigational Site Number : 8260005, Sutton, Surrey
  - Huddersfield Royal Infirmary - Investigational Site Number : 8260004, Huddersfield
  - Freeman Hospital - Investigational Site Number : 8260003, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org